CLINICAL TRIAL: NCT06436976
Title: The Effect of Probiotics ATG-F4 in Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chungnam National University Hospital (Other)
Collaborators: AtoGen Co. Ltd (Industry)
Responsible Party: Principal Investigator, Hyewon-Ryu, Professor, Chungnam National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CNUH 2023-08-012
Record Dates: First submitted 2024-02-18; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Cancer; Colon Cancer
Keywords: probiotics; pancreatic cancer; colon cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LT-002 (Lactobacillus reuteri ATG-F4) arm (Experimental): The group that will be consuming probiotics (LT-002 (Lactobacillus reuteri ATG-F4)) for 12 weeks. The subjects will take a daily intake of 4 x 10^10 colony forming unit (CFU) of LT-002.
  Interventions: Drug: LT-002 (Lactobacillus reuteri ATG-F4

INTERVENTIONS:
Drug: LT-002 (Lactobacillus reuteri ATG-F4 — The group that will be consuming probiotics for 12 weeks.

SUMMARY:
Patients with advanced colorectal cancer or pancreatic cancer who are receiving oxaliplatin-based chemotherapy will be included. The research participants in this study will consume probiotics along with safety and anti-cancer agent side effect-related questionnaires, blood, and fecal sample collection for up to 12 weeks from the date of registration. The total duration of participation for research subjects is 12 weeks.

DETAILED DESCRIPTION:
Chemotherapy is one of the cancer treatment methods, but some anticancer agents appear to influence the occurrence and progression of cachexia. Chemotherapy-Induced Cachexia refers to symptoms such as appetite loss, weight loss, muscle mass reduction, and fatigue caused by chemotherapy. While anticancer agents are used to eliminate or suppress tumor cells, most are administered intravenously, potentially causing damage not only to tumor cells but also to healthy cells and tissues. Cyclophosphamide, 5-fluorouracil (5-FU), and cisplatin induce negative nitrogen balance leading to weight loss, while cisplatin, irinotecan, adriamycin, and etoposide can cause muscle wasting through NF-κB activation. Additionally, muscle loss due to combination chemotherapy like FOLFIRI (5-fluorouracil, irinotecan, cisplatin) is associated with extracellular signal-regulated kinase 1/2 (ERK1/2) and p38 mitogen-activated protein kinase activation. Furthermore, research approached from a metabolic perspective has shown clear differences between cancer-induced cachexia and chemotherapy-induced cachexia, highlighting the need to differentiate and study cachexia induced by anticancer agents separately from cancer cachexia. In conclusion, while anticancer agents are essential for the demise of cancer cells and the inhibition of tumor growth, the occurrence of cachexia due to chemotherapy-induced damage to normal cells through prolonged administration poses a challenge that needs to be addressed to maintain the overall health of patients.

On the other hand, the microbiome refers to the total sum of all microorganisms present in a specific environment, and the human microbiome specifically refers to the collection of commensal, symbiotic, and pathogenic microorganisms coexisting with the human body. Approximately 95% of all microbes reside in the gastrointestinal tract, including the colon, and they are also widely distributed in the respiratory, reproductive, oral, and skin systems. The gut microbiome is known to play a crucial role in nutrient absorption, immune system regulation, and prevention of infectious diseases within the body.

Several studies suggest that changes in the composition and function of the gut microbiome may contribute to the development and progression of cachexia in cancer patients undergoing chemotherapy. In experiments where gut microbiota from mice treated with chemotherapy were transplanted into germ-free mice, an increase in inflammation-related C-X-C motif chemokine ligand 1 (CXCL1) was observed in the germ-free mice, accompanied by a significant decrease in their movement and physical activity. This result indicates that chemotherapy induces changes in the gut microbiota, which in turn can impact the entire body.

Chemotherapy can induce dysbiosis, an imbalance in the microbial community structure, leading to a reduction in beneficial bacteria and overgrowth of harmful bacteria, which can trigger inflammation and impair intestinal barrier function. Ultimately, this can promote inflammatory responses, exacerbating muscle loss and weight loss in cancer patients. Moreover, it can also affect nutrient absorption and metabolism, leading to malnutrition and energy imbalance.

Additionally, gut microbial communities produce various metabolites, such as short-chain fatty acids (SCFAs), which play important roles in host metabolism and immune function regulation. Dysbiosis may affect intestinal protein synthesis and energy metabolism. Overall, the profound involvement of the gut microbiome and metabolites in chemotherapy-induced cachexia symptoms suggests that microbiome-based therapies could be an interesting development target for alleviating or treating chemotherapy-induced cachexia.

Probiotics are generally known to improve gastrointestinal conditions such as constipation and diarrhea, inhibit harmful bacteria in the gut, and prevent diseases through their regulatory effects on intestinal function. They are also known to have effects such as immune enhancement, improvement of vaginal health, and alleviation of allergies. In particular, there is ongoing global research aimed at developing probiotics as therapeutic agents for the microbiome, which constitutes the total microorganisms in the gut. Recently, with the FDA approval of microbiome therapy for clostridiosis difficile infection, research in this area has been increasing.

The test strain of Lactobacillus reuteri ATG-F4 used in this study has been confirmed to be safe based on preclinical research results. When administered to mice transplanted with tumors and then treated with anticancer agents, it was observed to improve weight loss, muscle mass reduction, and muscle strength decline. Additionally, it helped alleviate diarrhea symptoms and normalize gut microbiota. These effects were found to be associated with the suppression of inflammatory responses induced by anticancer agents. Based on previous studies, this trial was planned to analyze the impact of the investigational product LT-002 (Lactobacillus reuteri ATG-F4) on the safety and improvement of anticancer agent side effects in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with advanced colorectal cancer or pancreatic cancer who are undergoing treatment with Oxaliplatin-based chemotherapy at Chungnam National University Hospital, including both newly diagnosed and recurrent cases.
* Aged 19 years or older.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2 points.
* Expected life expectancy of at least 3 months.
* Ability to understand the requirements of the clinical trial and willingness to sign the informed consent form.

Exclusion Criteria:

* Presence of known brain metastases.
* Malignant bowel obstruction requiring surgical intervention.
* Uncontrolled, active infections, symptomatic congestive heart failure, unstable angina, cardiac arrhythmias, or any psychiatric/social conditions that may limit compliance with the study requirements.
* Partial or complete intestinal obstruction.
* Pregnant or lactating women.
* Use of antibiotics, antifungals, or antiviral agents on more than one occasion within the past month.
* Consumption of probiotics products or fermented milk more than twice within the past month.
* Patients with neurological or psychiatric disorders.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of Body weight (Kg) | baseline, 4 weeks, 8 weeks
  Body weight measured by Bio-electrical Impedance Analysis

SECONDARY OUTCOMES:
Lean body mass | baseline, 4 weeks, 8 weeks
  Lean body mass measured by Bio-electrical Impedance Analysis
Body mass index | baseline, 4 weeks, 8 weeks
  kg/m^2
C-reactive protein | baseline, 4 weeks, 8 weeks
  C-reactive protein (mg/dL) measured by laboratory analysis
Interleukin-6 | baseline, 4 weeks, 8 weeks
  Interleukin-6 (pg/mL) measured by laboratory analysis
Neutrophil to lymphocyte ratio | baseline, 4 weeks, 8 weeks
  Absolute neutrophil count and lymphocyte count will be combined to report Neutrophil to lymphocyte ratio
Platelet to lymphocyte ratio | baseline, 4 weeks, 8 weeks
  Platelet and lymphocyte count will be combined to report Neutrophil to lymphocyte ratio
Progression-free survival | Up to 24 weeks, by 3 months
  Progression free survival (from initiation of chemotherapy to disease-progression or death, whenever occured first)
Overall survival | Up to 24 seeks, by 3 months
  Overall survival (from diagnosis to death)
effects of probiotics to Quality of life | baseline, 4 weeks, 8 weeks
  The EORTC Quality of life questionnaire - C30 score consists of 30 items divided into three subdomains: overall quality of life, functional areas, and symptom areas. Higher scores in the overall quality of life and functional areas indicate a better quality of life, while lower scores in the symptom areas also indicate a better quality of life.
Chemotherapy toxicity | baseline, 4 weeks, 8 weeks
  Chemotherapy toxicity Survey
Changes in gut microbiome profiles | baseline, 4 weeks, 8 weeks
  Changes in gut microbiome profiles, using 16s RNA analysis.
Hand grip strength | baseline, 4 weeks, 8 weeks
  Hand grip strength measurement using Digital grip strength dynamometer, T.K.K 5401, Japan). Hand grip strength will be measured to estimate the physical performances of participants.
Mid calf circumference | baseline, 4 weeks, 8 weeks
  Mid calf circumference will be measured to estimate the lean body mass of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Hyewon Ryu, Professor, Principal Investigator — Department of Hematology Oncology
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No
Due to the organization's policy, personal information of participants cannot be shared.